CLINICAL TRIAL: NCT03568747
Title: Efficacy and Mechanism of Non-invasive Ventilation in Relieving Dyspnea After Exercise in Patients With Stable Severe Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy and Mechanism of NIV in Relieving Dyspnea After Exercise in Patients With Stable Severe COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Yonger Ou, Principal Investigator, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GIRD201801
Record Dates: First submitted 2018-05-30; First posted 2018-06-26 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2018-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Noninvasive Ventilation; Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIV plus oxygen therapy (Experimental): noninvasive ventilation (dual-limb NIV) is given at peak exercise until the borg scale reaches it's baseline point
  Interventions: Device: noninvasive ventilation
- oxygen therapy (Experimental): oxygen therapy is given at peak exercise until the borg scale reaches it's baseline point
  Interventions: Device: oxygen therapy

INTERVENTIONS:
Device: noninvasive ventilation — dual-limb circuit NIV were given on maquet servo i apparatus
  Arms: NIV plus oxygen therapy
Device: oxygen therapy — oxygen therapy were introduced to the side port of the facemask
  Arms: oxygen therapy

SUMMARY:
Exertional dyspnea is a major cause of exercise limitation and anxiety, and contributes importantly to reduced quality of life for patients with COPD. The aim of this study is to determine the efficacy and mechanism of NIV with a dual-limb circuit plus oxygen therapy in relieving exertional dyspnea in patients with severe COPD, so as to provide a guidance for clinical use for NIV.

DETAILED DESCRIPTION:
Exertional dyspnea was the most characteristic respiratory symptoms in patients with chronic obstructive pulmonary disease (COPD), it is a major cause of exercise limitation and anxiety, and contributes importantly to reduced quality of life for patients with COPD. COPD patients often unconsciously adopt a sedentary lifestyle, probably due to distressing exertional dyspnea. The sedentarism results in physical deconditioning and alterations of the peripheral muscles, which leads to a vicious circle and contribute to the debilitation of the patients. Thereby, intervention should be taken to intervene this vicious cycle. It has been reported that noninvasive ventilation (NIV) could help unload the inspiratory muscle, improve dynamic pulmonary hyperinflation, improve neuro-mechanical coupling, oxygenation, and thus relieved dyspnea during exercise in COPD patients. However, in these reports, NIV was used as add-on therapy during exercise or at resting condition before exertional dyspnea occurred. So far, there's few studies on the efficacy of NIV used at the time of exertional dyspnea occurred as the rescue therapy to relieve dyspnea after exercise in patients with stable severe COPD while the patients are already undergoing optimal treatment with bronchodilator and anti-inflammatory medication, which might relieve their physiological and perceptional burden to limit their activities. The result of the investigators previous study has suggested that compared with oxygen therapy, NIV plus oxygen therapy resulted in decrease in dyspnea intensity at isotime, however, there's no statistically significant shortening in total dyspnea recovery time and NIV was not helpful in all the COPD patients. In another study, it was indicated that ventilated by a single-limb tubing with a plateau exhalation valve (PEV) caused CO2 rebreathing to COPD patients during exercise. CO2 rebreathing may have a negative impact on efficacy. Previous studies have proved that exercise tolerance was improved ventilated by noninvasive ventilation with a dual-limb circuit. In theory, NIV with a dual-limb circuit consists of one inhalation limb that introduces air into the patient's airways and one exhalation limb that leads exhaled gas outside of the airways, there is no risk of rebreathing. However, it is unclear whether NIV with a dual-limb circuit could be used at the time of exertional dyspnea occurred as rescue therapy to relieve dyspnea after exercise in patients with stable severe COPD and what are the mechanisms. The purpose of this study was therefore to determine whether assisted with NIV with dual-limb circuit in patients with stable severe COPD after exercise with exertional dyspnea (1)dyspnea was relieved after exercise in patients with stable severe COPD; (2)the repiratory mechanism.

ELIGIBILITY:
Inclusion Criteria:

* severe COPD (post bronchodilator FEV1/FVC < 70% and FEV1 < 50% predicted)
* stable clinical condition(no exacerbation in the 4 weeks prior to study participation with no change in medications)
* dyspnea as a main symptom that limited daily activities

Exclusion Criteria:

* obvious pulmonary bullae demonstrated by chest CT scan or X-ray examination facial trauma/malformation; recent facial, upper airway or upper gastrointestinal tract surgery
* systolic blood pressure > 160mmHg or diastolic blood pressure > 100mmHg at rest
* unstable angina or a myocardial infarct in the previous four weeks
* resting sinus tachycardia ( > 120 beats/min)
* patients with musculoskeletal or neurological disorders
* patients who are unable to give informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-23 (Actual); Primary Completion 2019-02-03 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
change from baseline Borg scale to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  this is a scale that asks the participants to rate the difficulty of breathing. It starts at number 0 where one's breathing is causing no difficulty at all and progresses through to number 10 where one's breathing difficulty is maximal.

SECONDARY OUTCOMES:
change from baseline diaphragm electromyogram to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  EMGdi
change from baseline index of neuromechanical dissociation of the respiratory system to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  EMGdi%max:Vt%VCpred

OTHER OUTCOMES:
change from baseline transdiaphragmatic pressure to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  Pdi
change from baseline esophageal pressure to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  Pes
change from baseline mouth pressure to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  Pm
change from baseline inspiratory capacity to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  IC
change from baseline minute ventilation to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  VE
change from baseline oxygen saturation to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  SpO2
change from baseline heart rate to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  HR
change from baseline total recovery time to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  total recovery time
change from baseline tidal volume to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  Vt
change from baseline respiratory rate to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  RR
change from baseline inspiratory time to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  Ti
change from baseline total duty cycle to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  Ttot
change from baseline expiratory time to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  Te
change from baseline pressure time product to complete recovery after exercise | baseline, at peak exercise and at every 30s interval until complete recovery
  PTP

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, Study Director — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China